CLINICAL TRIAL: NCT01585155
Title: Clinical Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of TA-650 in Pediatric Patients With Moderate to Severe Ulcerative Colitis.
Brief Title: Clinical Study of TA-650 in Pediatric Patients With Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TA-650-21
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Ulcerative Colitis
Keywords: Infliximab; REMICADE; TA-650
MeSH Terms: conditions — Pediatric ulcerative colitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TA-650 (Experimental)
  Interventions: Drug: TA-650

INTERVENTIONS:
Drug: TA-650 — TA-650 will be intravenously infused at 5 mg/kg as an induction regimen at Weeks 0, 2, 6. For subjects who meet the responder criteria, TA-650 will be administered at 8-week intervals thereafter until week 22.

SUMMARY:
The purpose of this study is to evaluate the the efficacy of TA-650 using Clinical activity index (CAI) score and other evaluation indicators in pediatric patients with moderate to severe ulcerative colitis after TA-650 administration of at a dose of 5 mg/kg at weeks 0, 2, and 6, and then every 8 weeks at weeks 14 and 22. The safety and pharmacokinetics are also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed as ulcerative colitis at least 3 months prior to screening.
* Have active ulcerative colitis despite adequate conventional therapy.

Exclusion Criteria:

* Patients who have severe pancolitis.
* Patients who have undergone surgery for ulcerative colitis within 8 weeks before enrollment or who were judged to require surgery for ulcerative colitis at enrollment.
* Patients who have a history of treatment with infliximab or other biologic products (anti-TNFα agents, anti-IL-6 agents, etc.).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2012-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toshifumi Hibi, MD, Study Director — Kitasato University Kitasato Institute Hospital; Kazuoki Kondo, MD, Study Director — Mitsubihsi Tanabe Pharma Corporation
Locations (7):
- Japan (7):
  - Investigational site, Chūbu
  - Investigational site, Hokkaido
  - Investigational site, Hokuriku
  - Investigational site, Kanto
  - Investigational site, Kinki
  - Investigational site, Kyusyu
  - Investigational site, Tōhoku

REFERENCES:
- [Result] Tajiri H, Arai K, Kagimoto S, Kunisaki R, Hida N, Sato N, Yamada H, Nagano M, Susuta Y, Ozaki K, Kondo K, Hibi T. Infliximab for pediatric patients with ulcerative colitis: a phase 3, open-label, uncontrolled, multicenter trial in Japan. BMC Pediatr. 2019 Oct 13;19(1):351. doi: 10.1186/s12887-019-1739-5. PMID 31607268

RESULTS

PARTICIPANT FLOW:
Groups:
- TA-650: Patients received TA-650 5 mg/kg at Weeks 0, 2, and 6; patients with a decreased CAI score at Week 8 were considered to be responders and received further doses at Week 14 and 22. Non-responders (patients with unchanged/increased CAI score) at Week 8 did not receive further study treatment. Assessments were conducted until Week 30 in responders and until Week 14 in non-responders.
Period: Overall Study
Arm/Group | TA-650
Started | 21
Completed | 16
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 2
Not completed — Worsening ulcerative colitis | 2

BASELINE CHARACTERISTICS:
Groups:
- TA-650: TA-650 is administered at a dose of 5 mg/kg at Weeks 0, 2 and 6, followed by administration at 8-week intervals at Weeks 14 and 22, based on the evaluation index such as CAI score.
Arm/Group | TA-650
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.7 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Who Achieved CAI Remission
Description: Clinical activity index (CAI) remission was defined as a case where a CAI score was not more than 4 on the evaluation day.
  CAI score was an activity index to evaluate disease activity, which is calculated as the sum (0 to 29 points) of subscores for 7 clinical conditions, consisting of the number of stools per week, blood in stools (based on weekly average), investigator's global assessment of the symptomatic state, abdominal pain/cramps, temperature elevation due to ulcerative colitis, extraintestinal manifestations, and laboratory findings (hemoglobin or ESR). A higher score indicates greater disease activity.
Time Frame: Weeks 2, 6, 8, 10, 14, 18, 22, 26, 30, and the last time point during the period from administration of the study drug to Week 30
Population: Five patients were discontinued. The reasons for discontinuation were adverse event in 1 patient, lack of efficacy in 2 patients, and worsening ulcerative colitis in 2 patients. Two non-responders were observed, and both of them completed the efficacy evaluation at Week 8.
Measure: Number; unit: percentage of participants
Arm/Group | TA-650
Number analyzed (Participants) | 21
percentage of participants
  Weeks 2: number analyzed (Participants) | 20
  Weeks 2 | 60.0
  Weeks 6: number analyzed (Participants) | 20
  Weeks 6 | 80.0
  Weeks 8: number analyzed (Participants) | 20
  Weeks 8 | 80.0
  Weeks 10: number analyzed (Participants) | 18
  Weeks 10 | 77.8
  Weeks 14: number analyzed (Participants) | 16
  Weeks 14 | 87.5
  Weeks 18: number analyzed (Participants) | 16
  Weeks 18 | 87.5
  Weeks 22: number analyzed (Participants) | 14
  Weeks 22 | 64.3
  Weeks 26: number analyzed (Participants) | 14
  Weeks 26 | 85.7
  Weeks 30: number analyzed (Participants) | 14
  Weeks 30 | 64.3
  The last time point | 42.9

2. Secondary Outcome: CAI Score
Description: CAI score was an activity index to evaluate disease activity, which is calculated as the sum (0 to 29 points) of subscores for 7 clinical conditions, consisting of the number of stools per week, blood in stools (based on weekly average), investigator's global assessment of the symptomatic state, abdominal pain/cramps, temperature elevation due to ulcerative colitis, extraintestinal manifestations, and laboratory findings (hemoglobin or ESR). A higher score indicates greater disease activity.
Time Frame: Baseline,Weeks 2, 6, 8, 10, 14, 18, 22, 26, 30, and the last time point during the period from administration of the study drug to Week 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TA-650
Number analyzed (Participants) | 21
units on a scale
  Baseline | 9.7 (2.7)
  Weeks 2: number analyzed (Participants) | 20
  Weeks 2 | 4.0 (3.2)
  Weeks 6: number analyzed (Participants) | 20
  Weeks 6 | 3.5 (3.5)
  Weeks 8: number analyzed (Participants) | 20
  Weeks 8 | 3.2 (3.5)
  Weeks 10: number analyzed (Participants) | 18
  Weeks 10 | 2.7 (2.9)
  Weeks 14: number analyzed (Participants) | 16
  Weeks 14 | 2.7 (3.0)
  Weeks 18: number analyzed (Participants) | 16
  Weeks 18 | 2.6 (2.6)
  Weeks 22: number analyzed (Participants) | 14
  Weeks 22 | 3.3 (3.1)
  Weeks 26: number analyzed (Participants) | 14
  Weeks 26 | 2.5 (2.3)
  Weeks 30: number analyzed (Participants) | 14
  Weeks 30 | 3.5 (2.2)
  The last time point | 5.6 (3.8)

3. Secondary Outcome: Partial Mayo Score
Description: Mayo score consists of four subscores (stool frequency, rectal bleeding, physician's global assessment and findings of endoscopy), each of which was assessed according to a four-level rating scale (0 to 3 points), and was determined from a total of the four subscores (0 to 12 points). In addition, the sum of the subscores (0 to 9 points) for stool frequency, rectal bleeding and physician's global assessment was used as a partial Mayo score. A higher score indicates greater disease activity.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TA-650
Number analyzed (Participants) | 21
units on a scale
  Baseline | 5.6 (1.6)
  Weeks 2: number analyzed (Participants) | 20
  Weeks 2 | 2.6 (2.3)
  Weeks 6: number analyzed (Participants) | 20
  Weeks 6 | 2.2 (2.0)
  Weeks 8: number analyzed (Participants) | 20
  Weeks 8 | 1.7 (1.7)
  Weeks 10: number analyzed (Participants) | 18
  Weeks 10 | 2.2 (2.1)
  Weeks 14: number analyzed (Participants) | 16
  Weeks 14 | 1.9 (1.9)
  Weeks 18: number analyzed (Participants) | 16
  Weeks 18 | 2.1 (1.8)
  Weeks 22: number analyzed (Participants) | 14
  Weeks 22 | 2.4 (2.1)
  Weeks 26: number analyzed (Participants) | 14
  Weeks 26 | 1.8 (1.7)
  Weeks 30: number analyzed (Participants) | 14
  Weeks 30 | 2.8 (1.9)
  The last time point | 3.7 (2.2)

4. Secondary Outcome: Pediatric Ulcerative Colitis Activity Index (PUCAI) Score
Description: PUCAI score was determined as a total of the subscores for each of the six evaluation items (0 to 85), including abdominal pain, rectal bleeding, stool consistency of most stools, number of stools per 24 hours, nocturnal stools and activity level. A higher score indicates greater disease activity.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TA-650
Number analyzed (Participants) | 21
units on a scale
  Baseline | 47.1 (15.2)
  Weeks 2: number analyzed (Participants) | 20
  Weeks 2 | 20.3 (16.3)
  Weeks 6: number analyzed (Participants) | 20
  Weeks 6 | 17.3 (17.5)
  Weeks 8: number analyzed (Participants) | 20
  Weeks 8 | 12.5 (13.5)
  Weeks 10: number analyzed (Participants) | 18
  Weeks 10 | 14.7 (16.9)
  Weeks 14: number analyzed (Participants) | 16
  Weeks 14 | 12.2 (12.0)
  Weeks 18: number analyzed (Participants) | 16
  Weeks 18 | 14.4 (16.8)
  Weeks 22: number analyzed (Participants) | 14
  Weeks 22 | 18.2 (15.6)
  Weeks 26: number analyzed (Participants) | 14
  Weeks 26 | 13.2 (14.0)
  Weeks 30: number analyzed (Participants) | 14
  Weeks 30 | 19.3 (18.8)
  The last time point | 28.8 (22.5)

ADVERSE EVENTS:
Arm/Group | TA-650
Serious Adverse Events (participants affected / at risk) | 3/21
Other Adverse Events (participants affected / at risk) | 19/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TA-650 (N=21)
Colitis ulcerative (Gastrointestinal disorders) | 2
Enterocolitis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TA-650 (N=21)
Bronchitis (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 7
Sinusitis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Anaemia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2
Headache (Nervous system disorders) | 1
Scleritis (Eye disorders) | 1
Vasculitis (Vascular disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Autoimmune pancreatitis (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Pancreatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Chest discomfort (General disorders) | 1
Infusion site pain (General disorders) | 1
Antinuclear antibody increased (Investigations) | 1
Blood pressure decreased (Investigations) | 1
Double stranded DNA antibody positive (Investigations) | 12
Protein urine present (Investigations) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other